CLINICAL TRIAL: NCT07195591
Title: Randomized Study of Resection and GammaTile® Followed by Concurrent External Beam Radiation Therapy (EBRT) and Temozolomide (TMZ) and Adjuvant TMZ Versus Standard of Care in Newly Diagnosed Glioblastoma (GBM)
Brief Title: Beginning Radiation Immediately With GammaTile at GBM Excision Versus Standard of Care
Acronym: BRIDGES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTM-105
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Newly Diagnosed; GammaTile; External Beam Radiation Therapy; Temozolomide; Brain; Tumor; Brachytherapy; Radiation Therapy; Surgery; Resection; GBM; BRIDGES; EBRT; TMZ
MeSH Terms: conditions — Glioblastoma; Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Maximal safe resection followed by EBRT with concurrent TMZ followed by adjuvant TMZ (Arm A) (Active Comparator): All patients will undergo tumor resection. Start TMZ (75 mg/m2/day orally) on the first day of EBRT and will be administered concurrently with EBRT, up to 5 days per week, for the 30-fraction course of EBRT for 6 weeks within 30±10 days post-surgery. After EBRT and concurrent TMZ phase, the first cycle begins 28 ±7 days following the last day of the EBRT and Concurrent TMZ Phase. Adjuvant TMZ includes 5 days of TMZ treatment at the start of each 28-day cycle. Additional cycles (up to a maximum of 12), which may be given at the discretion of the Investigator, will be documented, and performed in the same manner as done in the first 6 cycles.
  Interventions: Radiation: External Beam Radiation Therapy; Drug: Temozolomide
- Maximal safe resection + GammaTile followed by EBRT with concurrent TMZ then adjuvant TMZ (Arm B) (Experimental): All patients will undergo tumor resection + GammaTile implantation. Start TMZ (75 mg/m2/day orally) on the first day of EBRT and will be administered concurrently with EBRT, up to 5 days per week, for the 20-fraction course of EBRT for 4 weeks within 30±10 days post-surgery. After EBRT and concurrent TMZ phase, the first cycle begins 28 ±7 days following the last day of the EBRT and Concurrent TMZ Phase. Adjuvant TMZ includes 5 days of TMZ treatment at the start of each 28-day cycle. Additional cycles (up to a maximum of 12), which may be given at the discretion of the Investigator, will be documented, and performed in the same manner as done in the first 6 cycles.
  Interventions: Device: GammaTile®; Radiation: External Beam Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Device: GammaTile® — GammaTiles are a U.S. FDA-cleared, surgically targeted radiation therapy for patients with certain brain tumors. GammaTile consists of bioresorbable collagen tiles embedded with Cesium-131 (Cs-131) radioactive seeds
  Arms: Maximal safe resection + GammaTile followed by EBRT with concurrent TMZ then adjuvant TMZ (Arm B)
Radiation: External Beam Radiation Therapy — External beam radiation therapy (EBRT) is a type of radiation therapy that is standard of care. EBRT uses a machine outside the body to deliver high-energy beams of radiation to cancerous areas within the body
  Other Names: EBRT
Drug: Temozolomide — TMZ (Chemotherapy) is used as a first-line treatment, often in combination with radiation therapy after surgical resection of the tumor
  Other Names: TMZ

SUMMARY:
This is a Phase 3 prospective, randomized, superiority, open-label, multi-site study. The overview of this study is as follows:

* A Screening/Baseline Period of 21 days. During this time, patients will be randomized into a 1:2 allocation of Arm A:Arm B.
* A Perioperative/Operative Phase where patients will undergo tumor resection (Arm A) or tumor resection plus GammaTile implantation (Arm B).
* An EBRT Prior to Start Period. This occurs within 10 business days prior to EBRT and Concurrent TMZ Phase.
* An EBRT and Concurrent TMZ Phase, which will begin 30 ±10 days post-surgery. EBRT (30 fractions) and TMZ will be administered up to 5 days a week for 6 weeks in Arm A, and EBRT (20 fractions) and TMZ will be administered for up to 5 days a week for 4 weeks in Arm B. TMZ will be administered at a dose of 75 mg/m2/day orally for each Arm.
* An Adjuvant TMZ Phase, which begins 28 ±7 days following the EBRT and Concurrent TMZ Phase, and is comprised of six 28-day cycles. TMZ (150-200 mg/m2/day orally) will be administered for the first 5 days of each 28-day cycle for each Arm. Tumor treating fields are allowed but are not mandated during this phase. Up to 6 additional cycles (for a total of 12) can be completed at the discretion of the Investigator.
* An Early Discontinuation/Follow-Up Phase will occur 28 ±7 days after completion of Cycle 6 of the Adjuvant TMZ Phase, regardless of the total number of cycles completed or any delays in cycle start. If fewer than six cycles are completed, the first follow-up assessment will occur 28 ±7 days after the last administered dose of adjuvant TMZ. If patient has a qualifying event requiring entrance to Early Discontinuation Phase, the first follow-up assessment will occur as soon as feasible, but within 28 days.

For any unscheduled visits, data collected should be documented in the case report form (CRF) and must include, but are not limited to, safety evaluations, survival status, and disease status.

ELIGIBILITY:
Major Criteria Includes the Following:

Inclusion Criteria

* Patients must be ≥18 years of age.
* Have radiographic suspicion of newly diagnosed glioblastoma (GBM).

  o If final pathology reports IDH mutant glioma, then the patients found to have an IDH mutation will be followed for safety and QoL measures but will not be included in the primary and secondary comparative survival and efficacy analyses.
* Are medically and surgically appropriate for resection.
* Have an estimated Karnofsky Performance Scale (KPS) score of ≥70.
* Are able to receive standard of care treatment.

Exclusion Criteria

* A previous biopsy diagnosis other than IDH wild-type GBM.
* Have contraindications to TMZ, magnetic resonance imaging, gadolinium, or non-contrast computed tomography.
* Have multi-focal enhancing tumors that cannot be encompassed in one operative field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Days from surgery to death.
  The primary endpoint of the study is OS, defined as the day from surgery to death. Patients who are still alive (or lost to follow-up) at the time of data analysis will be censored at the last time point they were known to be alive.

SECONDARY OUTCOMES:
Progression Free Survival | Days from surgery to death or disease progression.
  To compare PFS, defined as days from surgery to death or disease progression, between the 2 study arms based on the most current RANO Resect Group criteria;
Time to next unplanned treatment | Time to next unplanned treatment.
  To compare the time to next unplanned treatment per study arm
Performance Status | 24 months.
  To assess the performance status up to 24 months
Safety Assessment | Study duration.
  To assess the nature, severity, and frequency of AEs between the 2 study arms based on the most current CTCAE criteria
Quality of Life Assessments | COST-Score duration of study; FACT-Br up to 12 months after randomization.
  Financial toxicity scale (Comprehensive Score for Financial Toxicity [COST]-score) and functional assessment of cancer therapy - brain (FACT-Br) up to 12 months after randomization.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Westchester Medical Center, Valhalla, New York
  - Brown University Health, Providence, Rhode Island